CLINICAL TRIAL: NCT06916039
Title: Randomized Controlled Nutrition Trial on Breakfast Glycaemic Index on the Course of Memory and Attention Among Young Adults - Relevance of Chronotype
Brief Title: Effects of Breakfast Glycaemic Index on Cognition in Earlier or Later Chronotypes.
Acronym: GlyCoBrainIn1
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anette Buyken (Other)
Collaborators: Paderborn University (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Anette Buyken, Anette Buyken, Paderborn University
Organization: Paderborn University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BU 1807/8-1-1
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: chronotype; breakfast; glycemic index; attention; cognition; memory; body composition; continous glucose monitoring; MCTQ

STUDY DESIGN:
Intervention Model Description: It is estimated that a maximum of 177 participants will need to be invited, to obtain full data sets from 44 participants of an earlier chronotype and 44 of a later chronotype each completing the cross-over designed intervention study. The intervention will consists of consumption of a carbohydrate-rich breakfast as a high-GI beverage at 8:40 p.m or a low-GI beverage at the same time. Participants will be randomly assigned to one of two groups stratified by chronotype: intake of a beverage with a high GI or low GI on day 1. On day 7, the meal of the high GI or low GI meal is switched. The trial is a two-arm cross-over study in which each participant serves as his / her own control to account for interindividual variations in diurnal glycaemic responses and cognitive performance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind, meaning that neither participants nor researchers know whether the consumed beverage has a high or low GI. Beverages will be pre-prepared by staff not involved in its provision.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high glycemic index breakfast (Experimental): 1. a high GI beverage (i.e. "glucose beverage") consisting of 75 g glucose dissolved in 500 ml tap water
  Interventions: Other: immediate verbal memory after high GI breakfast; Other: immediate verbal memory after low glycemic index breakfast
- low glycemic index breakfast (Experimental): 2. a low GI beverage inducing no reactive hypoglycaemia ("isomaltulose® beverage") consisting of 75 g isomaltulose dissolved in 500 ml tap water
  Interventions: Other: immediate verbal memory after high GI breakfast; Other: immediate verbal memory after low glycemic index breakfast

INTERVENTIONS:
Other: immediate verbal memory after high GI breakfast — Difference in immediate verbal memory after high GI breakfast at 150-180 minutes (i.e., in the late postprandial phase)
Other: immediate verbal memory after low glycemic index breakfast — Difference in immediate verbal memory after low GI breakfast at 150-180 minutes (i.e., in the late postprandial phase)

SUMMARY:
High glycaemic index (GI) breakfasts resulting in sharp rises in blood glucose may adversely affect memory and attention, particularly in the late postprandial phase (i.e., 120-180 minutes after breakfast). Previous research indicates that breakfast GI influences cognition in young adults, but many studies were too short to capture late postprandial effects. However, young adults may be particularly responsive to these adverse effects on cognition since they are prone to experience circadian misalignment in the morning due to the fact that their midpoint of sleep (i.e., chronotype) is biologically most delayed. Our recent research suggests that persons with later chronotypes do not display the known circadian decline in glucose tolerance as evidenced by equally high glycaemic responses to the identical high GI meal consumed in the morning or the evening. Hence, consuming an early breakfast "against the inner clock" may negatively affect glycaemic response particularly among persons with a later chronotype. Whether this vulnerability for persons with a later chronotype may extend to effects on cognition has not been examined.

Thus, the main objective of this controlled nutrition trial is to analyze the effects of a high versus a low GI beverage as a breakfast on subsequent memory and attention until 180 minutes after breakfast among young healthy university students. This will be examined in two samples, i.e. students with an earlier and with a later chronotype. Accordingly, our study will allow us to explore the relevance of chronotype for (i) the postprandial course of glucose levels and (ii) the course of memory and attention per se in the postprandial phase.

In preparation for the present study, at Paderborn University 356 students (aged 18-25) were enrolled between October 2024 and January 2025 in the GlyCoBrain Observational study (ID: NCT06679088) and were screened for their chronotypes. From these, persons with the earliest and latest chronotype will be invited to participate in the present cross-over designed study. It is planned that overall 88 persons will complete both intervention days consuming either a high GI or a low GI breakfast at 9:00 a.m. and undergoing repeated assessment of cognitive performance during the subsequent 180 minutes.

DETAILED DESCRIPTION:
Background Studies in young adults indicate beneficial effects of a low glycemic index (GI) breakfast on cognitive performance. A meta-analysis of 17 studies revealed benefits of a low-glycemic load (GL) breakfast on immediate memory only in the late post-prandial period. The meta-analysis reported no overall effect on attention in adults, yet suggests advantages for attention in children, adolescents, and young adults. A limitation of previous studies was that dairy was often allowed despite its strong insulinotropic effect, dampening the postprandial glycaemic response. To ensure an unbiased evaluation, the GlyCoBrain intervention study 1 will use pure water-carbohydrate mixtures, avoiding nutrient interactions, to examine the isolated effect of a high-GI breakfast.

Mechanisms explaining the time-dependent benefits of a low-GL breakfast are not fully understood. The provision of glucose to the brain is currently discussed as a central mechanism linking meal GI/GL to cognition. Generally, glucose is required for cognitive efforts as evidenced by decreases in local extracellular glucose concentrations in the activated brain area. The synthesis of key neurotransmitters in the brain requires a glucose supply. Glucose metabolism may be linked to memory via effects on tryptophan utilization and serotonin concentrations. Overall,the memory enhancing effect of glucose may require relatively constant blood glucose levels in the brain rather than high glucose amounts per se. Hence, whilst high GI foods elicit a transient increase in blood glucose level, low GI foods will result in a more sustained and longer-lasting provision of glucose. Since recent work suggests that there may be an optimal blood glucose range for cognitive performance and that this optimal range may differ by cognitive domain, it appears prudent to use continuous glucose monitoring in addition to the conventional measurement points directly before the cognitive test. However, benefits of low GI/GL breakfast for cognitive function have also been observed without differences in blood glucose levels. This may be attributable to an acutely improved postprandial insulin sensitivity and/or lower cortisol levels elicited by low GI meals. Accordingly, concomitant examinations of all three factors, i.e. glucose, insulin and cortisol levels, seem necessary to disentangle potential mechanisms.

The above mentioned meta-analysis also found greater benefits for individuals with better glucose tolerance, although this may be confounded by age. Studies suggest that young adults with poorer glucose tolerance, even within the healthy range, may be more vulnerable to these effects. While glucose tolerance follows a circadian rhythm, being lowest in the evening due to reduced pancreatic β-cell function and insulin response, circadian misalignment-common among young adults with later chronotypes-can also impair glucose tolerance, even at breakfast, due to decreased insulin sensitivity. This misalignment, often caused by social jetlag, has been linked to obesity, type 2 diabetes, and higher blood glucose and HbA1c levels, and an increased risk of depression. Considering results from our previous study showing high glucose responses among young adults with a late chronotype in the morning to a high GI breakfast, the GlyCoBrain intervention study 1 examines the hypothesis that consuming an early breakfast "against the inner clock" affects cognitive performance.

Hypothesis

(1) A low GI beverage breakfast (isomaltulose® beverage) results in a better memory and attention until 180 minutes compared to a high GI beverage breakfast (glucose beverage). (2) a low GI beverage breakfast results in fewer fluctuations in memory and attention throughout the morning. (3) the benefits of a low GI breakfast are particularly observed among people with later chronotype.

Aim The main objectives of this controlled nutrition trial are to analyze the effect of a high or low GI beverage at breakfast on memory and attention over the course of the morning including the late postprandial phase among young healthy university students. As young students are at high risk for a later chronotype, we aim to explore these effects in two samples of students with an earlier and later chronotype. In addition, our study will allow us to explore the relevance of chronotype for the postprandial course of glucose, insulin and cortisol levels.

Methodology Participants Healthy, German speaking students at Paderborn University with early or late chronotype.

Sample size calculation:

We base our sample size calculation on the difference in immediate memory and the study rated best in terms of quality in the meta-analysis. Given a standard deviation of 3.6 and 4.3 in both groups, and a standardized mean difference of 0.31 for people with a better glucose tolerance (corresponding to mean difference of 1.12) we require 44 participants in the smallest subgroup with a given power of 80% and alpha of 0.05 considering a correlation of 0.8 between both measurements (calculated with STATA, vers. 17.0). We assume, that 66% of invited students will participate and that 75% of those will complete the study. Hence, to have the full data set of 88 persons (44 with an early chronotype and 44 with a late chronotype) completing the trial, 117 need to start the trial and 177 people need to be invited from the GlyCoBrain Observational study which recruited 356 students from Paderborn University and screened for chronotype via MCTQ. In both chronotype samples equal sex distribution is envisaged.

Both samples will be invited to participate in the crossover nutrition trial, excluding smokers, people working on shift or having travelled for >2 time zone in the past 3 months, persons taking methylphenidate or using melatonin. Students will participate in 2 breakfast-cognition tests, each after an overnight fast at 8 a.m. to be taken over a course of 2 weeks including 1 week wash-out. Participants will randomly be assigned to one of two sequence groups, which differ only regarding the sequence of the intervention (Glucose beverage, isomaltulose® beverage or isomaltulose® beverage, glucose beverage). Randomization lists are provided by an external statistical advisor from the University of Esbjerg stratified by sex and chronotype. A randomized list was generated for 4 groups, each with 30 slots, using a block randomization approach. The randomization was performed using STATA (Vs 18.5; randomize) with 5 blocks, ensuring balance across the groups

Participants will receive to two different simple beverage breakfasts:

1. high GI beverage (glucose beverage) consisting of 75 g glucose dissolved in 500 ml tap water,
2. low GI beverage inducing no reactive hypoglycaemia (isomaltulose® beverage) consisting of 75 g isomaltulose dissolved in 500 ml tap water.

The intervention is structured into a 2-week schedule:

Week 1. Participants are invited for preparation day 1, during which a venous fasted blood sample is taken to determine fasting lipids, high-sensitivity-C-reactive protein, alanine aminotransferase and gamma-glutamyltransferase to metabolically characterize the recruited participants. To validate the consistency of the chronotype that had been determined in the GlyCoBrain Observational study previously, the participants' chronotype will again be determined via the Munich chronotype questionnaire. Body composition will be reassessed by Bioimpedance Analysis to estimate individual percentages of body fat, muscle mass, total body water and extracellular water. Additionally, body weight will be measured directly by the medical Body Composition Analyzer (mBCA, seca, Germany). Body height will be measured using an ultrasound measuring station (SECA287 db). Waist circumference will be assessed on the exposed upper body at the midpoint between the lower ribcage and the hip bone.

Continuous glucose monitoring (CGM, G7, Dexcom, Inc., San Diego,CA) is activated, accelerometry will be used to measure movement and sleep/wake conditions. A standardized evening meal will be provided to be consumed in the evening before the intervention to avoid secondary meal effects e.g. by pulse consumption. Participants will be asked to perform a training session on the cognition battery (see below).

The actual intervention starts three to five days later at 8 a.m. with each day running as follows:

* minimal invasive capillary blood samples collected at -40, 30, 80 and 140 minutes (in relation to the time point of drinking the beverage) will be used to determine glucose and insulin levels
* non-invasively cortisol samples from saliva at -40, 80 and 140 minutes
* continuous glucose measurements
* Heart rate belt to measure the heart rate variability in combination with the Unite fitness watch (Polar Electro, Finland).
* Cognition test at -30, 90 and 150 minutes
* test beverage breakfast including either Glucose or Isomaltulose to be drunken at time point 0, 9 a.m.
* appetite, thirst and mood will be assessed at -40, 30, 80 and 140 minutes each using a validated visual analogue scale
* removal of all devices and provision of a voluntary breakfast at 180 minutes Glucose levels will be directly determined using HemoCue Glucose 201 RT Analyzer (HemoCue AB, Schweden). Plasma insulin concentration and cortisol concentration in saliva will be determined by an enzyme-linked immunosorbent assay (ELISA) using a kit from IBL/Tecan.

Week 2. Again, participants repeat the preparation day as before (day 2), except for BIA, MCTQ and venous blood sample measurements. The intervention then continues 3 to 5 days after the preparation day following the same time scale as on intervention day 1.

Cognition tests Assessment using the test battery is expected to last approximately 25 minutes in total each time. Tests will include a set of tests developed by the ALA Institute Bochum, that was applied in our previous studies.

* verbal memory test (ability to correctly recall a total of 30 words immediately (recall) and after 20minutes (delayed recall))
* Visual-spatial short-term working memory test (Corsi-block tapping test equivalent, i.e., tapping a sequence of up to nine identical spatially separated blocks, sequentially increasing the difficulty by the number of presented blocks).
* Test of selective and sustained attention and visual scanning speed (modified version of the d2 Test of attention, during which the reaction specific signs within a series of presented signs will be assessed)
* Test of spatial attention and switching abilities between two different tasks (alternative version of the Trail Making Task)
* Test of tonic alertness (simple reaction time test).
* Test of inhibition, i.e. ability to inhibit a prepotent response, using a flanker task. In each trial three superposed triangles will be presented to the participants. The upper and lower triangles (flankers) will be pointing in the same direction but independent from the middle triangle (target). During the no-go trials a circle replaces the target. The participants will be supposed to press the buttons left or right according to the direction of the target or not to react in the case of a no-go condition. Each trial will be categorized as compatible-go, incompatible-go or no-go.
* A dummy test to ensure that delayed recall starts exactly 20 minutes after the immediate recall Statistical analysis Multilevel regression models will be used to analyze the effect of the interventions on verbal memory at 150-180 minutes. Identical models will be used for the other cognitive domains as outcome. Tests for interactions of the intervention effect with chronotype will be performed and stratified analyses by chronotype will be run. Note that consideration of interactions may also be relevant if p<0.1. Additional analyses will control for insulin sensitivity, cortisol, appetite, thirst and/or mood to explore whether observed effects may be partly attributable to these factors.

ELIGIBILITY:
Inclusion Criteria:

* Participants of GlyCoBrain Observational Study
* Early or late chronotype (approx. lowest and highest quartile)

Exclusion Criteria:

* Students studying nutritional science and home economics (study programs of the study PI)
* Intermediate chronotypes
* Persons unwilling to abstain from smoking or cannabis use during the intervention period
* Persons unwilling to consume standard evening meal prior to intervention days
* BMI>30 kg/m² (diurnal variation in glycaemic control is known to be absent among persons with obesity) and <18.5 kg/m2 (since underweight is also known to affect glucose homeostasis)
* acute or permanent use of sleep-promoting medications (including herbal preparation):

  * medications: melatonin, diphenhydramine, doxylamine
  * herbal preparations: hops, St. John's wort, lemon balm, lavender, passionflower, Baldurat, Neurexan, cannabinoids
* Use of psychotropic medications (antidepressants, tranquilizer, antipsychotics)
* Use of methylphenidate (e.g. Ritalin, Medikinet, Concerta)
* Use of cannabinoids by prescription
* Continuous administration of antihistamines when discontinuation is not feasible during the intervention
* Use of herbal preparations affecting memory and concentration (e.g. gingko, ginseng, ashwagandha)
* Use of other medications (e.g. insulin, metformin, SGLT2 inhibitors, steroids, ACE inhibitors)
* Selected chronic diseases (depression and other mental disorders such as anxiety disorder, ADHD, diabetes mellitus (all types), prediabetes, blood clotting disorders (e.g., thrombocytopenia, hemophilia), eating disorders (e.g., anorexia, binge eating, bulimia), Chronic inflammatory bowel diseases, infectious diseases (HIV, hepatitis), Addiction disorders (e.g., alcohol, drug, or medication dependency)
* Pregnant and breastfeeding individuals
* Shift work or travel in the past 3 months across more than 2 time zones
* students with a pacemaker/defibrillator or cochlear implant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in immediate verbal memory | 150-180 minutes
  Difference in immediate verbal memory between high and low GI breakfasts at 150-180 minutes (i.e., in the late postprandial phase)

CONTACTS AND LOCATIONS:
Overall Officials: Anette E Buyken, Prof. Dr., Principal Investigator — Paderborn University
Locations (1):
- Paderborn University, Paderborn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith MA, Riby LM, Eekelen JA, Foster JK. Glucose enhancement of human memory: a comprehensive research review of the glucose memory facilitation effect. Neurosci Biobehav Rev. 2011 Jan;35(3):770-83. doi: 10.1016/j.neubiorev.2010.09.008. Epub 2010 Sep 29. PMID 20883717
- [Background] Shrier I, Redelmeier A, Schnitzer ME, Steele RJ. Challenges in interpreting results from 'multiple regression' when there is interaction between covariates. BMJ Evid Based Med. 2021 Apr;26(2):53-56. doi: 10.1136/bmjebm-2019-111225. Epub 2019 Aug 22. PMID 31439540
- [Background] Schroder M, Muller K, Falkenstein M, Stehle P, Kersting M, Libuda L. Lunch at school and children's cognitive functioning in the early afternoon: results from the Cognition Intervention Study Dortmund Continued (CoCo). Br J Nutr. 2016 Oct;116(7):1298-1305. doi: 10.1017/S0007114516002932. Epub 2016 Sep 9. PMID 27608921
- [Background] Schroder M, Muller K, Falkenstein M, Stehle P, Kersting M, Libuda L. Short-term effects of lunch on children's executive cognitive functioning: The randomized crossover Cognition Intervention Study Dortmund PLUS (CogniDo PLUS). Physiol Behav. 2015 Dec 1;152(Pt A):307-14. doi: 10.1016/j.physbeh.2015.09.025. Epub 2015 Sep 30. PMID 26427889
- [Background] Sanchez-Aguadero N, Recio-Rodriguez JI, Patino-Alonso MC, Mora-Simon S, Alonso-Dominguez R, Sanchez-Salgado B, Gomez-Marcos MA, Garcia-Ortiz L. Postprandial effects of breakfast glycaemic index on cognitive performance among young, healthy adults: A crossover clinical trial. Nutr Neurosci. 2020 Jan;23(1):1-7. doi: 10.1080/1028415X.2018.1461459. Epub 2018 Apr 12. PMID 29649949
- [Background] Saad A, Dalla Man C, Nandy DK, Levine JA, Bharucha AE, Rizza RA, Basu R, Carter RE, Cobelli C, Kudva YC, Basu A. Diurnal pattern to insulin secretion and insulin action in healthy individuals. Diabetes. 2012 Nov;61(11):2691-700. doi: 10.2337/db11-1478. Epub 2012 Jun 29. PMID 22751690
- [Background] Philippou E, Constantinou M. The influence of glycemic index on cognitive functioning: a systematic review of the evidence. Adv Nutr. 2014 Mar 1;5(2):119-30. doi: 10.3945/an.113.004960. PMID 24618754
- [Background] Nabb SL, Benton D. The effect of the interaction between glucose tolerance and breakfasts varying in carbohydrate and fibre on mood and cognition. Nutr Neurosci. 2006 Jun-Aug;9(3-4):161-8. doi: 10.1080/10284150600955099. PMID 17176639
- [Background] Nabb S, Benton D. The influence on cognition of the interaction between the macro-nutrient content of breakfast and glucose tolerance. Physiol Behav. 2006 Jan 30;87(1):16-23. doi: 10.1016/j.physbeh.2005.08.034. Epub 2005 Oct 12. PMID 16225896
- [Background] Morris CJ, Yang JN, Garcia JI, Myers S, Bozzi I, Wang W, Buxton OM, Shea SA, Scheer FA. Endogenous circadian system and circadian misalignment impact glucose tolerance via separate mechanisms in humans. Proc Natl Acad Sci U S A. 2015 Apr 28;112(17):E2225-34. doi: 10.1073/pnas.1418955112. Epub 2015 Apr 13. PMID 25870289
- [Background] Lotti S, Pagliai G, Colombini B, Sofi F, Dinu M. Chronotype Differences in Energy Intake, Cardiometabolic Risk Parameters, Cancer, and Depression: A Systematic Review with Meta-Analysis of Observational Studies. Adv Nutr. 2022 Feb 1;13(1):269-281. doi: 10.1093/advances/nmab115. PMID 34549270
- [Background] Lamport DJ, Chadwick HK, Dye L, Mansfield MW, Lawton CL. A low glycaemic load breakfast can attenuate cognitive impairments observed in middle aged obese females with impaired glucose tolerance. Nutr Metab Cardiovasc Dis. 2014 Oct;24(10):1128-36. doi: 10.1016/j.numecd.2014.04.015. Epub 2014 May 14. PMID 24925124
- [Background] Kennedy DO, Scholey AB. Glucose administration, heart rate and cognitive performance: effects of increasing mental effort. Psychopharmacology (Berl). 2000 Mar;149(1):63-71. doi: 10.1007/s002139900335. PMID 10789884
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Dye L, Gilsenan MB, Quadt F, Martens VE, Bot A, Lasikiewicz N, Camidge D, Croden F, Lawton C. Manipulation of glycemic response with isomaltulose in a milk-based drink does not affect cognitive performance in healthy adults. Mol Nutr Food Res. 2010 Apr;54(4):506-15. doi: 10.1002/mnfr.200900196. PMID 20140897
- [Background] Donohoe RT, Benton D. Cognitive functioning is susceptible to the level of blood glucose. Psychopharmacology (Berl). 1999 Aug;145(4):378-85. doi: 10.1007/s002130051071. PMID 10460314
- [Background] Deng Q, Haszard JJ, Conner TS, Rapsey C, Peng M, Venn BJ. Cognitive performance, mood and satiety following ingestion of beverages imparting different glycaemic responses: a randomised double-blind crossover trial. Eur J Clin Nutr. 2021 Apr;75(4):602-610. doi: 10.1038/s41430-020-00749-6. Epub 2020 Sep 17. PMID 32943769
- [Background] Blaak EE, Antoine JM, Benton D, Bjorck I, Bozzetto L, Brouns F, Diamant M, Dye L, Hulshof T, Holst JJ, Lamport DJ, Laville M, Lawton CL, Meheust A, Nilson A, Normand S, Rivellese AA, Theis S, Torekov SS, Vinoy S. Impact of postprandial glycaemia on health and prevention of disease. Obes Rev. 2012 Oct;13(10):923-84. doi: 10.1111/j.1467-789X.2012.01011.x. Epub 2012 Jul 11. PMID 22780564
- [Background] Benton D, Ruffin MP, Lassel T, Nabb S, Messaoudi M, Vinoy S, Desor D, Lang V. The delivery rate of dietary carbohydrates affects cognitive performance in both rats and humans. Psychopharmacology (Berl). 2003 Feb;166(1):86-90. doi: 10.1007/s00213-002-1334-5. Epub 2002 Dec 12. PMID 12488949
- [Background] Benton D, Nabb S. Breakfasts that release glucose at different speeds interact with previous alcohol intake to influence cognition and mood before and after lunch. Behav Neurosci. 2004 Oct;118(5):936-43. doi: 10.1037/0735-7044.118.5.936. PMID 15506876
- [Background] Anderson JR, Hawkins MAW, Updegraff J, Gunstad J, Spitznagel MB. Baseline glucoregulatory function moderates the effect of dairy milk and fruit juice on postprandial cognition in healthy young adults. Eur J Nutr. 2018 Oct;57(7):2343-2352. doi: 10.1007/s00394-017-1505-0. Epub 2017 Jul 13. PMID 28707217
- [Background] Anderson JR, Maki KC, Palacios OM, Edirisinghe I, Burton-Freeman B, Spitznagel MB. Varying roles of glucoregulatory function measures in postprandial cognition following milk consumption. Eur J Nutr. 2021 Apr;60(3):1499-1510. doi: 10.1007/s00394-020-02343-9. Epub 2020 Jul 31. PMID 32737613
- [Background] Gaylor CM, Benton D, Brennan A, Young HA. The impact of glycaemic load on cognitive performance: A meta-analysis and guiding principles for future research. Neurosci Biobehav Rev. 2022 Oct;141:104824. doi: 10.1016/j.neubiorev.2022.104824. Epub 2022 Aug 11. PMID 35963545